CLINICAL TRIAL: NCT04364737
Title: CONTAIN COVID-19: Convalescent Plasma to Limit Coronavirus Associated Complications: a Randomized Blinded Phase 2 Study Comparing the Efficacy and Safety of Anti-SARS-CoV2 Plasma to Placebo in COVID-19 Hospitalized Patients
Brief Title: CONTAIN COVID-19: Convalescent Plasma to Limit COVID-19 Complications in Hospitalized Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Albert Einstein College of Medicine (Other); Yale University (Other); The University of Texas Health Science Center, Houston (Other); The University of Texas Health Science Center at Tyler (Other); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-00541
Record Dates: First submitted 2020-04-22; First posted 2020-04-28 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Coronavirus; Coronavirus Infection
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent donor plasma (Active Comparator)
  Interventions: Biological: Convalescent Plasma
- Lactated ringer's solution or sterile saline solution (Placebo Comparator)
  Interventions: Other: Saline solution

INTERVENTIONS:
Biological: Convalescent Plasma — SARS-CoV-2 convalescent plasma (1-2 units; ~250-500 mL) with antibodies to SARS-CoV-21 per April 13, 2020 directive by the FDA, obtained from New York Blood Center will be administered to eligible candidate
  Arms: Convalescent donor plasma
Other: Saline solution — Equivalent volume of saline solution (defined as half-,quarter-, or normal saline) will be administered to eligible candidate as a placebo control group.
  Arms: Lactated ringer's solution or sterile saline solution

SUMMARY:
This is a randomized, blinded phase 2 trial that will assess the efficacy and safety of anti-SARS-CoV-2 convalescent plasma in hospitalized patients with acute respiratory symptoms requiring oxygen supplementation.

DETAILED DESCRIPTION:
A total of 300 eligible subjects will be randomized in a 1:1 ratio to receive either convalescent plasma (CP) from people who have recovered from COVID-19 containing antibodies to SARS-CoV-2 or a placebo control, Lactated Ringer's Solution (LR) or saline solution (SS). Hospitalized COVID-19 patients aged ≥18 years of age with respiratory symptoms within 3 to 7 days from the onset of illness OR within 3 days of hospitalization will be eligible to participate.

ELIGIBILITY:
Inclusion Criteria

1. Patients ≥18 years of age
2. Hospitalized with laboratory confirmed COVID-19
3. One or more of the following respiratory signs or symptoms: cough, chest pain, shortness of breath, fever, oxygen saturation ≤ 94%, abnormal CXR/CT imaging)
4. Hospitalized for ≤ 72 hours OR within day 3 to 7 days from first signs of illness
5. On supplemental oxygen, non-invasive ventilation or high-flow oxygen
6. Patients may be on other randomized controlled trials of pharmaceuticals for COVID -19 and patients who meet eligibility criteria will not be excluded on this basis.

Exclusion Criteria

1. Receipt of pooled immunoglobulin in past 30 days
2. Contraindication to transfusion or history of prior reactions to transfusion blood products
3. Invasive mechanical ventilation or extracorporeal membrane oxygenation (ECMO)
4. Volume overload secondary to congestive heart failure or renal failure
5. Unlikely to survive past 72 hours from screening based on the assessment of the investigator
6. Unlikely to be able to assess and follow outcome due to poor functional status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 941 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2022-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mila B Ortigoza, MD, PhD, Principal Investigator — NYU Langone Health
Locations (9):
- United States (9):
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Miami Hospital and Clinics, Miami, Florida
  - NYU Langone Health, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - University of Texas Rio Grande Valley, Edinburg, Texas
  - The University of Texas Health Science Center, Houston, Texas
  - The University of Texas Health Science Center, Tyler, Texas
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin / Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie the results reported in this article, after deidenficiation (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to Mila.Ortigoza@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Ortigoza MB, Yoon H, Goldfeld KS, Troxel AB, Daily JP, Wu Y, Li Y, Wu D, Cobb GF, Baptiste G, O'Keeffe M, Corpuz MO, Ostrosky-Zeichner L, Amin A, Zacharioudakis IM, Jayaweera DT, Wu Y, Philley JV, Devine MS, Desruisseaux MS, Santin AD, Anjan S, Mathew R, Patel B, Nigo M, Upadhyay R, Kupferman T, Dentino AN, Nanchal R, Merlo CA, Hager DN, Chandran K, Lai JR, Rivera J, Bikash CR, Lasso G, Hilbert TP, Paroder M, Asencio AA, Liu M, Petkova E, Bragat A, Shaker R, McPherson DD, Sacco RL, Keller MJ, Grudzen CR, Hochman JS, Pirofski LA; CONTAIN COVID-19 Consortium for the CONTAIN COVID-19 Study Group; Parameswaran L, Corcoran AT, Rohatgi A, Wronska MW, Wu X, Srinivasan R, Deng FM, Filardo TD, Pendse J, Blaser SB, Whyte O, Gallagher JM, Thomas OE, Ramos D, Sturm-Reganato CL, Fong CC, Daus IM, Payoen AG, Chiofolo JT, Friedman MT, Wu DW, Jacobson JL, Schneider JG, Sarwar UN, Wang HE, Huebinger RM, Dronavalli G, Bai Y, Grimes CZ, Eldin KW, Umana VE, Martin JG, Heath TR, Bello FO, Ransford DL, Laurent-Rolle M, Shenoi SV, Akide-Ndunge OB, Thapa B, Peterson JL, Knauf K, Patel SU, Cheney LL, Tormey CA, Hendrickson JE. Efficacy and Safety of COVID-19 Convalescent Plasma in Hospitalized Patients: A Randomized Clinical Trial. JAMA Intern Med. 2022 Feb 1;182(2):115-126. doi: 10.1001/jamainternmed.2021.6850. PMID 34901997

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Convalescent Donor Plasma | Lactated Ringer's Solution or Sterile Saline Solution
Started | 468 | 473
Completed | 463 | 463
Not Completed | 5 | 10
Not completed — Withdrawal by Subject | 4 | 9
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Donor Plasma | Lactated Ringer's Solution or Sterile Saline Solution | Total
Number analyzed (Participants) | 463 | 463 | 926
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (15.2) | 63.3 (15.1) | 62.35 (15.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 197 | 381
  Male | 279 | 266 | 545
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 181 | 186 | 367
  Not Hispanic or Latino | 282 | 277 | 559
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 41 | 30 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 68 | 139
  White | 256 | 278 | 534
  More than one race | 76 | 70 | 146
  Unknown or Not Reported | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 463 | 463 | 926

OUTCOME MEASURES:

1. Primary Outcome: Score on the WHO 11-point Ordinal Scale for Clinical Improvement at 14 Days
Description: Uninfected 0 Uninfected; no viral RNA detected Ambulatory 1 Asymptomatic; viral RNA detected 2 Symptomatic; Independent 3 Symptomatic; assistance needed
  Hospitalized:
  Mild disease 4 Hospitalized; no oxygen therapy 5 Hospitalized; oxygen by mask or nasal prongs
  Hospitalized:
  Severe disease 6 Hospitalized; oxygen by NIV or High flow 7 Intubation & Mechanical ventilation; pO2/FIO2 >/= 150 or SpO2/FIO2 >/=200 8 Mechanical ventilation pO2/FIO2 < 150 (SpO2/FIO2 <200) or vasopressors 9 Mechanical ventilation pO2/FIO2 < 150 and vasopressors, dialysis or ECMO Death 10 Dead
Time Frame: 14 days post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Convalescent Donor Plasma | Lactated Ringer's Solution or Sterile Saline Solution
Number analyzed (Participants) | 463 | 463
score on a scale | 2 [2 to 5] | 2 [2 to 5]

2. Secondary Outcome: Score on the WHO 11-point Ordinal Scale for Clinical Improvement at 28 Days
Description: as for outcome 1
Time Frame: 28 days post-randomization
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Convalescent Donor Plasma | Lactated Ringer's Solution or Sterile Saline Solution
Number analyzed (Participants) | 462 | 462
score on a scale | 2 [1 to 3] | 2 [1 to 4]

ADVERSE EVENTS:
Time Frame: 90 days from baseline
Description: Regular investigator assessment at baseline, days 1, 3, 7, 14, 28, 60, and 90.
Arm/Group | Convalescent Donor Plasma | Lactated Ringer's Solution or Sterile Saline Solution
All-Cause Mortality (participants affected / at risk) | 4/468 | 3/473
Serious Adverse Events (participants affected / at risk) | 112/468 | 108/473
Other Adverse Events (participants affected / at risk) | 147/468 | 136/473
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Donor Plasma (N=468) | Lactated Ringer's Solution or Sterile Saline Solution (N=473)
Abdominal wall haematoma (Gastrointestinal disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 16 | 19
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 9 | 8
Atrial fibrillation (Cardiac disorders) | 14 | 7
Bacteraemia (Infections and infestations) | 3 | 11
Bradycardia (Cardiac disorders) | 0 | 2
Candida pneumonia (Infections and infestations) | 0 | 2
Cardiac arrest (Cardiac disorders) | 61 | 70
Cerebral infarction (Nervous system disorders) | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 2 | 0
Chest pain (General disorders) | 4 | 3
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Coronavirus test positive (Investigations) | 0 | 2
Cytomegalovirus viraemia (Infections and infestations) | 2 | 2
Death (General disorders) | 4 | 3
Deep vein thrombosis (Vascular disorders) | 12 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Embolic stroke (Nervous system disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Fall (Injury, poisoning and procedural complications) | 3 | 0
Fibrin D dimer increased (Investigations) | 4 | 8
Fungaemia (Infections and infestations) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 11 | 4
Haematoma (Vascular disorders) | 0 | 4
Haematuria (Renal and urinary disorders) | 2 | 0
Haemorrhage (Vascular disorders) | 0 | 2
Haemorrhagic stroke (Nervous system disorders) | 0 | 2
Hepatic enzyme increased (Investigations) | 5 | 3
Hospice care (Surgical and medical procedures) | 11 | 12
Hospitalisation (Surgical and medical procedures) | 2 | 0
Hypotension (Vascular disorders) | 38 | 55
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 69 | 56
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 2
Liver function test increased (Investigations) | 3 | 4
Lung assist device therapy (Surgical and medical procedures) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 9 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pneumonia (Infections and infestations) | 3 | 0
Pneumonia bacterial (Infections and infestations) | 15 | 24
Pneumonia klebsiella (Infections and infestations) | 2 | 3
Pneumonia pseudomonal (Infections and infestations) | 4 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Pulmonary haemorrhage (Vascular disorders) | 2 | 0
Renal failure (Renal and urinary disorders) | 17 | 23
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 65 | 76
Retroperitoneal haematoma (Vascular disorders) | 0 | 2
Sepsis (Infections and infestations) | 0 | 5
Staphylococcal bacteraemia (Infections and infestations) | 3 | 3
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 2
Supraventricular tachycardia (Cardiac disorders) | 5 | 7
Systemic candida (Infections and infestations) | 2 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 0
Tracheostomy (Surgical and medical procedures) | 4 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Urinary tract infection (Infections and infestations) | 7 | 11
Ventricular fibrillation (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Donor Plasma (N=468) | Lactated Ringer's Solution or Sterile Saline Solution (N=473)
Acute kidney injury (Renal and urinary disorders) | 23 | 16
Alanine aminotransferase increased (Investigations) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 10 | 8
Aspartate aminotransferase increase (Investigations) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 12 | 7
Bacteraemia (Infections and infestations) | 2 | 2
Cardiac arrest (Cardiac disorders) | 2 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
C-reactive protein increased (Investigations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 9 | 8
Delivery (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Enterococcal bacteraemia (Infections and infestations) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Fibrin D dimer increased (Investigations) | 4 | 3
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Haematoma (Vascular disorders) | 2 | 0
Hepatic enzyme increased (Investigations) | 8 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Hypotension (Vascular disorders) | 8 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Leukocytosis (Blood and lymphatic system disorders) | 3 | 5
Liver function test increased (Investigations) | 10 | 11
Oral candidiasis (Infections and infestations) | 2 | 2
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 4 | 2
Pneumonia klebsiella (Infections and infestations) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 5
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Transfusion reaction (Injury, poisoning and procedural complications) | 3 | 0
Transaminases increased (Investigations) | 0 | 2
Troponin increased (Investigations) | 0 | 4
Troponin T increased (Investigations) | 2 | 0
Urinary tract infection (Infections and infestations) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT04364737/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-28): https://cdn.clinicaltrials.gov/large-docs/37/NCT04364737/ICF_000.pdf